CLINICAL TRIAL: NCT02425332
Title: Validation of Lokomat-aided Assessment of Gait Ability
Brief Title: Validation of a Novel Robot-aided Assessment of Gait Ability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: KEK-ZH-2015 0020/PB_2016-00466
Record Dates: First submitted 2015-04-20; First posted 2015-04-23 (Estimated); Last update posted 2017-12-19 (Actual); Status verified 2017-12

CONDITIONS: Spinal Cord Injury
Keywords: Spinal Cord Injury; adaptive control; assessment; assist-as-needed; walking ability; Lokomat
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lokomat assessment (Experimental)
  Interventions: Device: Lokomat gait trainer

INTERVENTIONS:
Device: Lokomat gait trainer

SUMMARY:
The aim of this study is the validation of a novel gait assessment method implemented in the Lokomat gait trainer with respect to established clinical gait assessment methods. The walking assessment method is based on the progressive reduction of the support of the device. The outcome measures of this algorithm will be the support needed in the different gait phases (guidance force of hip and knee joints) and the support required to the body weight support system (unloading). The hypothesis is that the guidance force and the support of the device will converge to a profile individual for each subject that is representative of one's impairment in the different gait phases. The reliability of the method will be tested collecting data from two sessions of Lokomat training. The validity of the method will be tested comparing the outcome of the assessment task with established clinical walking assessment measures.

ELIGIBILITY:
Inclusion Criteria:

* individuals >1 year post Spinal Cord Injury or able bodied persons

Exclusion Criteria:

* presence of contraindications to Lokomat training, inability or unwillingness to provide written informed consent or follow study procedures

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-05; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Intraclass Correlation Coefficient between Lokomat score. | up to one week
  Reliability of Lokomat assessment

CONTACTS AND LOCATIONS:
Locations (1):
- Universitätsklinik Balgrist, Zurich, Switzerland

REFERENCES:
- [Derived] Maggioni S, Lunenburger L, Riener R, Curt A, Bolliger M, Melendez-Calderon A. Assessing walking ability using a robotic gait trainer: opportunities and limitations of assist-as-needed control in spinal cord injury. J Neuroeng Rehabil. 2023 Sep 21;20(1):121. doi: 10.1186/s12984-023-01226-4. PMID 37735690